CLINICAL TRIAL: NCT05580029
Title: Open Label Prospective Trial of Fractional Ablative CO 2 Resurfacing With Laser- Facilitated Steroid Delivery in Patients With Mild to Moderate Hidradenitis Suppurativa.
Brief Title: Fractional CO2 Laser Fenestration and Steroid Delivery in HS Lesions
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Timothy Gillenwater, Principal Investigator, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APP-22-04651
Record Dates: First submitted 2022-09-30; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Scar; Hidradenitis Suppurativa
MeSH Terms: conditions — Cicatrix; Hidradenitis Suppurativa | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Intervention Model Description: Hurley stage I or stage II disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Triamcinolone Topical — The treatments will consist of fractional ablative CO2 laser therapies followed by topical application of triamcinolone dosed at 40 mg/ml.
Procedure: Fractional Ablative CO2 Therapy — 1st pass: 30-40 mJ at 5% density. 2nd pass: 120 mJ at 1% density
Drug: EMLA 5% cream — 2 g/10cm2 Topical 30 minutes before each fractional ablative CO2 session

SUMMARY:
Assess the efficacy of fractional ablative CO2 therapy combined with topical steroids in HS patients with Hurley stage I or stage II disease.

Hidradenitis suppurativa (HS) is a chronic, oftentimes debilitating inflammatory skin condition that presents with painful lesions in intertriginous areas of the body. The reported prevalence of HS in the U.S. is around 1-4%. Medical therapies, which typically consist of topical or systemic antibiotics, hormone- regulating drugs, and immunomodulators, are initially used to control the disease but HS can be recalcitrant to these modalities in the long-term. Optimizing management of mild-moderate HS is crucial to prevent disease progression and improve patients' quality of life.

DETAILED DESCRIPTION:
This is an open label prospective study aimed at understanding the efficacy of fractional ablative CO 2 laser therapy combined with steroids in HS patients with mild-moderate (Hurley stage I or stage II) disease. Study subjects will be patients with mild-moderate HS. The subjects will undergo a minimum of 3 treatment sessions and up to 5 treatment sessions at 4-6 week intervals. Patients will be informed of the aim of the study and the risks and benefits of the intervention. All questions that the subjects have will be answered and patients will be informed that their participation is completely voluntary. Subjects who agree and consent to participate in the study will partake in the treatment sessions. EMLA™ 5% cream will be applied as a topical anesthetic to the affected area 30 minutes prior to treatment. Fractional ablative CO 2 laser therapy will be performed and the HS lesions that will be treated include: non-inflammatory and inflammatory nodules, sinus tracts, abscesses, and scars. The fractional CO 2 laser treatment will be followed by immediate application of triamcinolone acetonide 40 mg/ml to the treatment area. Patients will be evaluated before the 1st treatment session and before every subsequent treatment session. The last study visit will occur 1 month after the completion of the last treatment session. Before each laser treatment, physicians will perform a complete assessment of Hurley stage and HS-PGA score. The number of non-inflammatory nodules, inflammatory nodules, abscesses, and sinus tracts in the treated area will be counted. Patients will evaluate their pain and itch level and provide their impression on whether their HS has improved, worsened, or stayed the same. Patients will also complete the Patient Global Assessment Item questionnaire. For scars, objective scar assessment will be performed using the Fibrometer ® , Elastimeter ® , and SkinColorCatch ® measurement tools. The Fibrometer ® measures tissue induration and skin stiffness. The Elastimeter ® induces constant skin deformation and returns a measurement of skin elasticity. The SkinColorCatch ® is a colorimeter that allows skin tone to be measured. Measurements of scars will be taken before each treatment session. In addition, the scars will be assessed using the VSS and POSAS scales by the investigators. Patients will also complete a POSAS self- assessment at each treatment session. Pictures of the treatment area will be taken during each visit with permission from the patients to analyze the effects of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older with a diagnosis of HS for at least 6 months
* Subjects who provide informed consent to undergo the procedure
* Patients with mild to moderate HS (Hurley stage I or stage II)
* Must not have been using topical or systemic therapies for 2 weeks prior to starting treatment on the affected area
* The use of antiseptic washes and intralesional steroid injections for acute lesions (rescue therapy) will be allowed

Exclusion Criteria:

* Under the age of 18
* Pregnant women
* Severe HS (Hurley stage III)
* Using topical or systemic medications within the 2 weeks prior to starting therapy
* History of adverse reactions to laser resurfacing or steroids
* Other diseases besides HS which require ongoing systemic therapies
* Active infection within the treatment area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-01-20 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Endpoint Measure of non-inflammatory nodules | After each treatment session (4-6 weeks)
  Change from baseline in number of non-inflammatory nodules
Endpoint measure of Fibrometer measurements | Before and after each treatment session (4-6 weeks)
  Change in Fibrometer® measurements
Endpoint Measure of Elastimeter | Before and after each treatment session (4-6 weeks)
  Change in Elastimeter®
Endpoint measure of self-reported improvement in HS | After each treatment session (4-6 weeks)
  Proportion of patients who self-report improvement in HS
Endpoint measure of inflammatory nodules | After each treatment session (4-6 weeks)
  Change from baseline in number of inflammatory nodules
Endpoint measure in SkinColorCatch | Before and after each treatment session (4-6 weeks)
  Change in SkinColorCatch® measurements
Endpoint measure of sinus tracts | After each treatment session (4-6 weeks)
  Change from baseline in number of sinus tracts
Endpoint measure of abscesses | After each treatment session (4-6 weeks)
  Change from baseline in number of abscesses
Endpoint measure of pain/itch level | After each treatment session (4-6 weeks)
  Change from baseline in pain/itch levels Scaled (1-10)
Endpoint measure in investigator assessed VSS score | Before and after each treatment session (4-6 weeks)
  Change in investigator assessed VSS
  Vancouver scar scale :
  Vascularity : normal, pink, red, purple (0-3) Pigmentation : normal, hypopigmentation, hyperpigmentation (0-2) Pliability : normal, supple, yielding, firm, banding, contracture (0-5) Height: normal (flat), 0-2mm, 2-5mm, >5mm (0-3)
Endpoint Measure in investigator assessed POSAS score | Before and after each treatment session (4-6 weeks)
  Change in investigator assessed POSAS scores Vascularity (0-10) Pigmentation (0-10) Thickness (0-10) Relief (0-10) Pliability (0-10) Surface area (0-10) Overall opinion (0-10)
Endpoint measure of HS-PGA scores | After each treatment session (4-6 weeks)
  Change from baseline in HS-PGA scores Scaled (0-5)
Endpoint measure in patient assessed POSAS score | Before and after each treatment session (4-6 weeks)
  Change in patient assessed POSAS score
Endpoint measure of changes in patient global assessment questionnaire scores | After each treatment session (4-6 weeks)
  Change from baseline in Patient Global Assessment questionnaire scores

REFERENCES:
- [Result] Alikhan A, Lynch PJ, Eisen DB. Hidradenitis suppurativa: a comprehensive review. J Am Acad Dermatol. 2009 Apr;60(4):539-61; quiz 562-3. doi: 10.1016/j.jaad.2008.11.911. PMID 19293006
- [Result] Jemec GB. Clinical practice. Hidradenitis suppurativa. N Engl J Med. 2012 Jan 12;366(2):158-64. doi: 10.1056/NEJMcp1014163. No abstract available. PMID 22236226
- [Result] Goldburg SR, Strober BE, Payette MJ. Hidradenitis suppurativa: Epidemiology, clinical presentation, and pathogenesis. J Am Acad Dermatol. 2020 May;82(5):1045-1058. doi: 10.1016/j.jaad.2019.08.090. Epub 2019 Oct 9. PMID 31604104
- [Result] Preda-Naumescu A, Ahmed HN, Mayo TT, Yusuf N. Hidradenitis suppurativa: pathogenesis, clinical presentation, epidemiology, and comorbid associations. Int J Dermatol. 2021 Nov;60(11):e449-e458. doi: 10.1111/ijd.15579. Epub 2021 Apr 22. PMID 33890304
- [Result] Ring HC, Riis Mikkelsen P, Miller IM, Jenssen H, Fuursted K, Saunte DM, Jemec GB. The bacteriology of hidradenitis suppurativa: a systematic review. Exp Dermatol. 2015 Oct;24(10):727-31. doi: 10.1111/exd.12793. Epub 2015 Aug 21. PMID 26119625
- [Result] Nguyen TV, Damiani G, Orenstein LAV, Hamzavi I, Jemec GB. Hidradenitis suppurativa: an update on epidemiology, phenotypes, diagnosis, pathogenesis, comorbidities and quality of life. J Eur Acad Dermatol Venereol. 2021 Jan;35(1):50-61. doi: 10.1111/jdv.16677. Epub 2020 Jul 16. PMID 32460374
- [Result] Worden A, Yoho DJ, Houin H, Moquin K, Hamzavi I, Saab I, Siddiqui A. Factors Affecting Healing in the Treatment of Hidradenitis Suppurativa. Ann Plast Surg. 2020 Apr;84(4):436-440. doi: 10.1097/SAP.0000000000002105. PMID 31688123
- [Result] Alikhan A, Sayed C, Alavi A, Alhusayen R, Brassard A, Burkhart C, Crowell K, Eisen DB, Gottlieb AB, Hamzavi I, Hazen PG, Jaleel T, Kimball AB, Kirby J, Lowes MA, Micheletti R, Miller A, Naik HB, Orgill D, Poulin Y. North American clinical management guidelines for hidradenitis suppurativa: A publication from the United States and Canadian Hidradenitis Suppurativa Foundations: Part I: Diagnosis, evaluation, and the use of complementary and procedural management. J Am Acad Dermatol. 2019 Jul;81(1):76-90. doi: 10.1016/j.jaad.2019.02.067. Epub 2019 Mar 11. PMID 30872156
- [Result] Hamzavi IH, Griffith JL, Riyaz F, Hessam S, Bechara FG. Laser and light-based treatment options for hidradenitis suppurativa. J Am Acad Dermatol. 2015 Nov;73(5 Suppl 1):S78-81. doi: 10.1016/j.jaad.2015.07.050. PMID 26470622
- [Result] Das K, Daveluy S, Kroumpouzos G, Agarwal K, Podder I, Farnbach K, Ortega-Loayza AG, Szepietowski JC, Grabbe S, Goldust M. Efficacy and Toxicity of Classical Immunosuppressants, Retinoids and Biologics in Hidradenitis Suppurativa. J Clin Med. 2022 Jan 27;11(3):670. doi: 10.3390/jcm11030670. PMID 35160122
- [Result] Lapins J, Sartorius K, Emtestam L. Scanner-assisted carbon dioxide laser surgery: a retrospective follow-up study of patients with hidradenitis suppurativa. J Am Acad Dermatol. 2002 Aug;47(2):280-5. doi: 10.1067/mjd.2002.124601. PMID 12140476
- [Result] Madan V, Hindle E, Hussain W, August PJ. Outcomes of treatment of nine cases of recalcitrant severe hidradenitis suppurativa with carbon dioxide laser. Br J Dermatol. 2008 Dec;159(6):1309-14. doi: 10.1111/j.1365-2133.2008.08932.x. PMID 19036028
- [Result] Hazen PG, Hazen BP. Hidradenitis suppurativa: successful treatment using carbon dioxide laser excision and marsupialization. Dermatol Surg. 2010 Feb;36(2):208-13. doi: 10.1111/j.1524-4725.2009.01427.x. Epub 2009 Dec 21. PMID 20039918
- [Result] Ramsdell WM. Fractional carbon dioxide laser resurfacing. Semin Plast Surg. 2012 Aug;26(3):125-30. doi: 10.1055/s-0032-1329414. PMID 23904820
- [Result] Tierney E, Mahmoud BH, Hexsel C, Ozog D, Hamzavi I. Randomized control trial for the treatment of hidradenitis suppurativa with a neodymium-doped yttrium aluminium garnet laser. Dermatol Surg. 2009 Aug;35(8):1188-98. doi: 10.1111/j.1524-4725.2009.01214.x. Epub 2009 May 12. PMID 19438670
- [Result] Riis PT, Boer J, Prens EP, Saunte DM, Deckers IE, Emtestam L, Sartorius K, Jemec GB. Intralesional triamcinolone for flares of hidradenitis suppurativa (HS): A case series. J Am Acad Dermatol. 2016 Dec;75(6):1151-1155. doi: 10.1016/j.jaad.2016.06.049. Epub 2016 Sep 28. PMID 27692735
- [Result] Wang J, Wu J, Xu M, Gao Q, Chen B, Wang F, Song H. Combination therapy of refractory keloid with ultrapulse fractional carbon dioxide (CO2 ) laser and topical triamcinolone in Asians-long-term prevention of keloid recurrence. Dermatol Ther. 2020 Nov;33(6):e14359. doi: 10.1111/dth.14359. Epub 2020 Oct 12. PMID 33002270
- [Result] Waibel JS, Wulkan AJ, Shumaker PR. Treatment of hypertrophic scars using laser and laser assisted corticosteroid delivery. Lasers Surg Med. 2013 Mar;45(3):135-40. doi: 10.1002/lsm.22120. Epub 2013 Mar 4. PMID 23460557
- [Result] Alakad R, Nassar A, Atef H, Eldeeb F. Fractional CO2 Laser-Assisted Delivery Versus Intralesional Injection of Methotrexate in Psoriatic Nails. Dermatol Surg. 2022 May 1;48(5):539-544. doi: 10.1097/DSS.0000000000003418. Epub 2022 Mar 24. PMID 35333217
- [Result] Majid I, Jeelani S, Imran S. Fractional Carbon Dioxide Laser in Combination with Topical Corticosteroid Application in Resistant Alopecia Areata: A Case Series. J Cutan Aesthet Surg. 2018 Oct-Dec;11(4):217-221. doi: 10.4103/JCAS.JCAS_96_18. PMID 30886476
- [Result] Haedersdal M, Sakamoto FH, Farinelli WA, Doukas AG, Tam J, Anderson RR. Fractional CO(2) laser-assisted drug delivery. Lasers Surg Med. 2010 Feb;42(2):113-22. doi: 10.1002/lsm.20860. PMID 20166154
- [Result] Morelli Coppola M, Salzillo R, Segreto F, Persichetti P. Triamcinolone acetonide intralesional injection for the treatment of keloid scars: patient selection and perspectives. Clin Cosmet Investig Dermatol. 2018 Jul 24;11:387-396. doi: 10.2147/CCID.S133672. eCollection 2018. PMID 30087573
- [Result] Coondoo A, Phiske M, Verma S, Lahiri K. Side-effects of topical steroids: A long overdue revisit. Indian Dermatol Online J. 2014 Oct;5(4):416-25. doi: 10.4103/2229-5178.142483. PMID 25396122